CLINICAL TRIAL: NCT03379766
Title: Quality Control of CE-Certified Phonak Hearing Aids - 2017_37
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Sonova2017_37
Record Dates: First submitted 2017-12-13; First posted 2017-12-20 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Successor of Phonak Audéo B-Direct (Experimental): The successor of Phonak Audéo B-Direct will be fitted to the participants individual hearing loss.
  Interventions: Device: Successor of Phonak Audéo B-Direct
- Phonak Audéo B-Direct (Active Comparator): The Phonak Audéo B-Direct will be fitted to the participants individual hearing loss.
  Interventions: Device: Phonak Audéo B-Direct

INTERVENTIONS:
Device: Successor of Phonak Audéo B-Direct — The successor of Phonak Audéo B-Direct will be fitted to the participants indivudal hearing loss.
  Arms: Successor of Phonak Audéo B-Direct
Device: Phonak Audéo B-Direct — The Phonak Audéo B-Direct will be fitted to the participants individual hearing loss.
  Arms: Phonak Audéo B-Direct

SUMMARY:
Phonak Hearing Systems pass through different development and study stages. At an early stage, feasibility studies are conducted to investigate new algorithms, features and functions in an isolated manner. If the benefit is proven, their performance is then investigated regarding interdependency between all available algorithms, features and functions running in parallel in a hearing aid (pivotal/pre-validation studies) and, as a result, they get optimized. Afterwards, and prior to product launch, the Phonak Hearing Systems undergo a final quality control in terms of clinical trials. This is a pre-validation study, investigating optimized algorithms, features and functions. This will be a clinical evaluation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Adult hearing impaired persons (minimum age: 18 years) with at least 3 months experience with hearing aids
* Good written and spoken (Swiss) German language skills
* Healthy outer ear
* Ability to fill in a questionnaire (p/eCRF) conscientiously
* Informed Consent as documented by signature

Exclusion Criteria:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments in Stäfa (Switzerland)
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Central hearing disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Spontaneous acceptance of the initial pre-calculation (first fit) | One week
  The data, serving as primary outcomes are collected in the first study appointment. The spontaneous acceptance of the initial pre-calculation (also called 'first fit') in regard to loudness and sound quality will be assessed with the aid of a systematic interview in lab.

SECONDARY OUTCOMES:
Listening effort in noisy listening environment | One week
  The data, serving as secondary outcomes are collected in the second study appointment. The listening effort in noisy listening environments will be assessed under controlled conditions in lab with the aid of the Adaptive Categorial Listening Effort Scaling Test (ACALES). The result shows the listening effort on a scale from 'no effort - extreme effort' at different signal to noise ratios.
Speech intelligibility in noisy listening environment | One week
  The data, serving as secondary outcomes are collected in the third study appointment. The speech intelligibility in noise will be assessed with the aid of the german Oldenburg sentence test (OLSA) under controlled conditions in lab. The result is the signal to noise ratio in dB (dB SNR).

OTHER OUTCOMES:
TV streaming | Three weeks
  The data, serving as other outcomes are collected within home trials with the test hearing aids, which take place between the weekly study appointments. The participants will be asked to assess the streamed signals in regard to any disturbing artefacts (e. g. fluctuation of volume or sound quality). In case that the participants experienced such artefacts, they will be asked to rate how bothersome these artefacts were (on a 10-point scale from 'not at all - extremely'). These ratings will be aggregated to arrive at one reported value.

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No